CLINICAL TRIAL: NCT04495049
Title: Vivity Insight: A Study of Patient Satisfaction and Visual Performance
Status: Completed | Type: Observational
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 1911 Vivity ALC57290333
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2020-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Alcon Vivity or Vivity Toric IOL — Patients who previously underwent cataract surgery with the Alcon Vivity or Vivity Toric IOL in both eyes.

SUMMARY:
This will be a single arm, open-label, prospective study of patient-reported outcomes of patients with bilateral implantation of the Vivity or Vivity Toric implant.

DETAILED DESCRIPTION:
Existing diffractive extended depth of focus (EDOF) lenses provide two adjacent "zones" of uncorrected vision (distance and intermediate or intermediate and near) but have a track record of frequent patient dissatisfaction because of unwanted visual side effects, "spider webs" or haloes. The Vivity non-diffractive EDOF lens offers this same range ofvision with contrast sensitivity similar to a monofocal lens, which suggests fewer side effects will be encountered in clinical practice.

This study is designed to measure postoperative patient-reported outcomes with this new lens implant. Previous studies we have conducted on the bilateral ReSTOR 3.0, ReSTOR with ActiveFocus 2.5 (mixed with 3.0 and alone with mini-monovision) have shown high satisfaction, spectacle independence, and acceptable glare and halo profiles using a validated questionnaire instrument developed by MDbackline, Inc. The postoperative portions of this study will be designed to mirror those previous studies using the same instrument.

All subjects will receive the Vivity or Vivity Toric implant binocularly with a target of plano sphere.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract and otherwise healthy eyes, not exhibiting any significant ocular morbidity that would be expected to influence outcome measures.
* Patients implanted with Vivity or Vivity Toric lenses bilaterally within 6 months of the survey administration.
* Patients whose postoperative manifest refraction at the time of the survey is within ± 0.5 D sphere and ≤0.75 D of cylindrical refraction.
* Patients who have given consent to participate in the survey.

Exclusion Criteria:

* Patients with visually significant co-morbidities (corneal, retina, optic nerve disease) that could affect their satisfaction with surgery.
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered IOL, cystoid macular edema, etc.) that would, the judgement of the investigator, influence the outcome measures of the study.
* Patients with previous refractive surgery within the past 6 months prior to cataract surgery.
* Patients with > grade 1 posterior capsule opacity at their last visit.
* Patients who do not meet the refractive endpoints described in the Inclusion Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cataract surgery.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reporting "not at all" or "just a little" when asked, "With or without glasses, how much do you notice glare or haloes around lights in dim light situations?" | 8/1/2020 - 7/1/2021
  Percentage of patients reporting "not at all" or "just a little" when asked, "With or without glasses, how much do you notice glare or haloes around lights in dim light situations?"

SECONDARY OUTCOMES:
Percentage of postoperative patients who report "rarely" when asked "How often do you need glasses to see the computer?" | 8/1/2020 - 7/1/2021
  Percentage of postoperative patients who report "rarely" when asked "How often do you need glasses to see the computer?"
Percentage of postoperative patients who report that they do not require reading glasses for various activities | 8/1/2020 - 7/1/2021
  Percentage of postoperative patients who report that they do not require reading glasses for various activities (driving, reading, including fine print, seeing computer monitor, watching TV, sports/hobbies when asked "For what types of activities do you need glasses to see (other than sunglasses)?"

OTHER OUTCOMES:
Percentage of patients reporting "very satisfied" when asked, "Overall, how satisfied are you with your vision after your latest surgery?" | 8/1/2020 - 7/1/2021
  Percentage of patients reporting "very satisfied" when asked, "Overall, how satisfied are you with your vision after your latest surgery?"
Percentage of patients who report "very satisfied" or "satisfied" to the same question. | 8/1/2020 - 7/1/2021
  Percentage of patients who report "very satisfied" or "satisfied" to the same question.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Harvard Eye Associates, Laguna Hills, California
  - Quentin Allen, Palm City, Florida
  - Quantum Vision Center, Edwardsville, Illinois